CLINICAL TRIAL: NCT00007085
Title: Prospective Investigation of Pulmonary Embolism Diagnosis (PIOPED II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Diagnostic
Other Study IDs: 132; U01HL063942 (NIH)
Record Dates: First submitted 2000-12-07; First posted 2000-12-08 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Lung Diseases; Pulmonary Embolism; Venous Thromboembolism
MeSH Terms: conditions — Lung Diseases; Pulmonary Embolism; Venous Thromboembolism | interventions — Tomography, X-Ray Computed

INTERVENTIONS:
Device: Tomography, X-ray Computed

SUMMARY:
To determine the value of contrast enhanced spiral computed tomography (spiral CT) for the diagnosis of acute pulmonary embolism (PE).

DETAILED DESCRIPTION:
BACKGROUND:

Approximately 600,000 Americans sustain pulmonary embolism each year; one-third of these episodes are fatal. Unfortunately, pulmonary embolism is underdiagnosed and, therefore, under-treated. A substantial body of evidence suggests that the diagnosis of pulmonary embolism is not made in the majority of patients in whom it causes or contributes to death.

In the main, there are two explanations for the failure to diagnose pulmonary embolism: pulmonary embolism may be clinically silent, and there is no definitive, noninvasive diagnostic test. Indeed, ventilation perfusion lung scans are nondiagnostic in the majority of patients with suspected acute pulmonary embolism. Pulmonary angiography may be used to establish a diagnosis in such patients, but it is underutilized because of a mortality risk around 1 percent.

Recently, relatively small studies have suggested that contrast enhanced spiral computed tomography (CT) scanning is a useful diagnostic test for pulmonary embolism, with sensitivity as high as 80 percent and specificity as high as 95 percent. Spiral CT is widely available and much less invasive than pulmonary angiography. If spiral CT could be established as a useful diagnostic test, pulmonary embolism would be diagnosed more effectively and more patients would receive proper treatment.

DESIGN NARRATIVE:

The study evaluates the role of spiral CT scan in the diagnosis of PE by comparison with a composite reference test, including pulmonary angiography, V/Q lung scan in patients without prior PE and compression ultrasound of the lower extremities in patients with no prior deep venous thrombosis (DVT).

ELIGIBILITY:
> 18% normal kidney function, no dye allergies, suspected of acute pulmonary embolism

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fowler — George Washington University; Charles Hales — Massachusetts General Hospital; Russell Hull — University of Calgary; Kenneth Leeper — Emory University; John Popovich — Case Western Reserve Univ-Henry Ford HSC; Henry Sostman — Weill Medical College of Cornell University; Paul Stein — St. Joseph Mercy; Victor Tapson — Duke University; John Weg — University of Michigan at Ann Arbor; Pamela Woodard — Washington University School of Medicine

REFERENCES:
- [Background] Gottschalk A, Stein PD, Goodman LR, Sostman HD. Overview of Prospective Investigation of Pulmonary Embolism Diagnosis II. Semin Nucl Med. 2002 Jul;32(3):173-82. doi: 10.1053/snuc.2002.124177. PMID 12105798